CLINICAL TRIAL: NCT01214954
Title: Early Rehabilitation After Toal Hip Replacement. -Effect of Supervised Progressive Resistance Training
Brief Title: Early Rehabilitation After Total Hip Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Regionshospitalet Silkeborg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M-20090231
Record Dates: First submitted 2010-09-17; First posted 2010-10-05 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Osteoarthritis, Hip
Keywords: Total Hip Replacement; Rehabilitation; Resistance training
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Active Comparator): Standard rehabilitation
  Interventions: Other: Control group
- Resistance training (Experimental): 10 weeks of supervised progressive resistance training initiated within the first week after total hip replacement.
  Interventions: Other: Supervised progressive resistance training

INTERVENTIONS:
Other: Supervised progressive resistance training — Resistance training 2 times/week initiated within the first week after total hip replacement. The training is supervised by physiotherapists and individually progressed.
  Arms: Resistance training
Other: Control group — Standard rehabilitation consisting of home-based exercises with 2 postoperative instructions by a physiotherapist.
  Arms: Control group

SUMMARY:
The purpose of this study is to determine whether supervised progressive resistance training is effective in the early phase after Total Hip Replacement. The investigators hypothesise that 10 weeks of supervised, progressive resistance training immediately after discharge will lead to increased functional performance, muscle strength and muscle power compared to standard rehabilitation consisting of home-based exercise.

DETAILED DESCRIPTION:
After total hip replacement (THR) surgery there is a documented deficit in muscle strength and functional performance. There is a lack of evidence concerning the effectiveness of postoperative physiotherapy and training, however a few small studies have shown promising effect of resistance training.

The present study will provide new and important knowledge concerning the effect of different rehabilitation strategies after THR. This might lead to a change in the rehabilitation regimes and faster and better recovery after THR surgery.

ELIGIBILITY:
Inclusion Criteria:

* Total hip replacement for osteoarthrosis
* Living within 30 km from the hospital
* Motivated to attend training 2 times/week in 10 weeks
* Reduced functional ability measured as: HOOS score < 67
* written informed consent

Exclusion Criteria:

* Comorbidities such as cancer, neuromuscular diseases, heart diseases etc.
* Cognitive impairment
* Body mass index > 35
* Resurfacing prosthesis
* Scheduled additional prosthetic surgery in lower extremity within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2010-09; Primary Completion 2013-01 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Leg extension power | 10 weeks postoperative
  The power in leg extension is measured using the Nottingham leg extension power rig. Data is provided in watt and adjusted for bodyweight (watt/kg)

SECONDARY OUTCOMES:
Walking speed | 4 weeks postoperative
  Maximal walking speed measured over 20 m.
Sit-to-stand | 10 weeks postoperative
  The maximal number of rises from a chair within 30 seconds
Stair test | 10 weeks postoperative
  The time taken to ascend 18 steps as fast as possible
Hip Osteoarthritis Outcome Score (HOOS) | 6 months postoperative
  Questionnaire. A disease-specific patient reported outcome measure of function, pain, sport/recreation and quality of life related to the hip.
Walking speed | 10 weeks
  Maximal walking speed measured over 20 m.
Walking speed | 6 months postoperative
  Maximal walking speed measured over 20 m.
Leg extension power | 6 months postoperative
  The power in leg extension is measured using the Nottingham leg extension power rig. Data is provided in watt and adjusted for bodyweight (watt/kg)
Sit-to-stand | 6 months postoperative
  The maximal number of rises from a chair within 30 seconds
Stair test | 6 months postoperative
  The time taken to ascend 18 steps as fast as possible
Hip Osteoarthritis Outcome Score (HOOS) | 2 weeks postoperative
  Questionnaire. A disease-specific patient reported outcome measure of function, pain, sport/recreation and quality of life related to the hip.
Hip Osteoarthritis Outcome Score (HOOS) | 4 weeks postoperative
  Questionnaire. A disease-specific patient reported outcome measure of function, pain, sport/recreation and quality of life related to the hip.
Hip Osteoarthritis Outcome Score (HOOS) | 6 weeks postoperative
  Questionnaire. A disease-specific patient reported outcome measure of function, pain, sport/recreation and quality of life related to the hip.
Isometric muscle strength | 4 weeks postoperative
  Test of isometric muscle strength in hip abduction and hip flexion using hand-held dynamometry
Isometric muscle strength | 10 weeks postoperative
  Test of isometric muscle strength in hip abduction and hip flexion using hand-held dynamometry
Isometric muscle strength | 6 months postoperative
  Test of isometric muscle strength in hip abduction and hip flexion using hand-held dynamometry
Gait quality | 10 weeks postoperative
  Instrumented gait analysis using a combined accelerometer and gyro-sensor in 20 meter walk test and stair climb test. The purpose is to measure asymmetry between limps during walking and stair climbing and compare the two groups according to these variables. This outcome measure is performed on a subgroup of participants (n=26, 13 in each group)
Gait quality | 6 months postoperative
  Instrumented gait analysis using a combined accelerometer and gyro-sensor in 20 meter walk test and stair climb test. The purpose is to measure asymmetry between limps during walking and stair climbing and compare the two groups according to these variables. This outcome measure is performed on a subgroup of participants (n=26, 13 in each group)
Hip Osteoarthritis Outcome Score (HOOS) | 10 weeks postoperative
  Questionnaire. A disease-specific patient reported outcome measure of function, pain, sport/recreation and quality of life related to the hip.
Hip Osteoarthritis Outcome Score (HOOS) | 1 year postoperative
  Questionnaire. A disease-specific patient reported outcome measure of function, pain, sport/recreation and quality of life related to the hip.

CONTACTS AND LOCATIONS:
Overall Officials: Lone R Mikkelsen, MSc., Principal Investigator — University of Aarhus
Locations (1):
- Silkeborg Regional Hospital, Silkeborg, Denmark

REFERENCES:
- [Derived] Mikkelsen LR, Petersen AK, Mechlenburg I, Mikkelsen S, Soballe K, Bandholm T. Description of load progression and pain response during progressive resistance training early after total hip arthroplasty: secondary analyses from a randomized controlled trial. Clin Rehabil. 2017 Jan;31(1):11-22. doi: 10.1177/0269215516628305. Epub 2016 Jul 10. PMID 26851251
- [Derived] Mikkelsen LR, Mechlenburg I, Soballe K, Jorgensen LB, Mikkelsen S, Bandholm T, Petersen AK. Effect of early supervised progressive resistance training compared to unsupervised home-based exercise after fast-track total hip replacement applied to patients with preoperative functional limitations. A single-blinded randomised controlled trial. Osteoarthritis Cartilage. 2014 Dec;22(12):2051-8. doi: 10.1016/j.joca.2014.09.025. Epub 2014 Oct 22. PMID 25305374